CLINICAL TRIAL: NCT04139213
Title: Comparing Medication Maintenance in Comprehensive Community and Pharmacy Settings to Enhance Engagement
Brief Title: Medication Maintenance Therapy in Community Pharmacy Settings
Acronym: MATPharm
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lifespan (Other)
Collaborators: University of Rhode Island (Other); The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Traci Green, Senior Research Scientist, Lifespan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9919
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination; vivitrol; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (Active Comparator): usual medication assisted treatment for maintenance care of opioid use disorder
  Interventions: Drug: buprenorphine/naloxone oral product; Drug: injectable naltrexone; Drug: oral naltrexone
- Pharmacy MAT (Experimental): pharmacy-based medication assisted treatment for maintenance care of opioid use disorder
  Interventions: Drug: buprenorphine/naloxone oral product; Drug: injectable naltrexone; Other: Pharmacy maintenance addiction care; Drug: oral naltrexone

INTERVENTIONS:
Drug: buprenorphine/naloxone oral product — To treat opioid use disorder, buprenorphine/naloxone will be provided by a study pharmacist under a collaborative pharmacy practice agreement on a weekly or monthly basis, unless the care plan specifies greater frequency of pharmacy visit. The median expected dose of buprenorphine/naloxone (sublingual film or tablet) is 8 to 24 mg daily, and may be adjusted per the collaborative pharmacy practice agreement.
  Other Names: Suboxone
Drug: injectable naltrexone — To treat opioid use disorder, injectable naltrexone will be provided by a study pharmacist under a collaborative pharmacy practice agreement on a monthly (injectable naltrexone) basis. The expected dose of injectable naltrexone will be approximately 380 mg. Injectable naltrexone will be dispensed and prepared by the pharmacist but administered by nursing staff for the pilot study.
  Other Names: Vivitrol
Other: Pharmacy maintenance addiction care — Patients randomized to the pharmacy study arm and on a stable dose of buprenorphine/naloxone or naltrexone will receive maintenance care at the pharmacy for up to three months. Patients will visit for check-ins with a pharmacist on a monthly, weekly, or more frequent basis, depending on the individual treatment plan. Patients on buprenorphine/naloxone will be dispensed their medication at study visits, whereas patients taking injectable naltrexone will be dispensed it monthly by the pharmacist. All patients will visit the pharmacy at least monthly for addiction care (assessment, toxicological testing).
  Arms: Pharmacy MAT
Drug: oral naltrexone — To augment care for patients receiving injectable naltrexone for the treatment of OUD and treat cravings that may arise before their scheduled injection, patients prescribed injectable naltrexone may be provided a several day supply of oral naltrexone by a study pharmacist under a collaborative pharmacy practice agreement. The expected dose of oral naltrexone will be approximately 25-50 mg daily.

SUMMARY:
The goal of this study is to compare pharmacy-based medication assisted treatment (MAT) with usual care MAT for people with opioid use disorder.

DETAILED DESCRIPTION:
This study compares pharmacy-based medication assisted treatment (MAT) with usual care MAT. This will be the first study to use a randomized controlled trial design to test the multisite implementation of known effective interventions to treat opioid use disorder and prevent fatal opioid overdose (treatment with buprenorphine and natlrexone) in a community pharmacy setting. Understanding how this model can improve engagement in care within innovative systems of MAT delivery like the Rhode Island Centers of Excellence in MAT model as well as the more traditional office based opioid therapy (OBOT) arrangement, and for patients with shorter and longer time on stabilized MAT doses advances the science of addiction health services.

This study presents an opportunity to compare clinical outcomes of patients randomized to receive the same medications but in different settings that are equipped with differing levels of counseling expectations and access to wrap-around services. In this way, the trial helps to inform whether-and for whom--the limited support services in the pharmacy are sufficient to engage and retain patients in MAT, or if ready access to comprehensive services are necessary. Approximately 86% of Americans live within 5 miles of a pharmacy, making pharmacists the most accessible health care professionals. This model could redefine the role of the pharmacy.

The completed initial phase of the study (Phase 1) involved a pilot of the pharmacy MAT care model. The current phase of the study (Phase 2) is a randomized controlled trial comparing the pharmacy MAT care model to usual MAT care.

The aim of the current phase is to conduct a randomized controlled trial of 250 medication-stabilized (with BNX or NTX) patients with OUD receiving MAT care in Rhode Island, comparing engagement and clinical outcomes for patients followed up in a usual care model to those maintained and followed up in a pharmacy MAT care model.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English speaking
* Currently enrolled at a MAT site for the treatment of OUD, maintained on a stable MAT (BNX, NTX) dose for at least 2 days or interested in induction
* Able and willing to provide written informed consent and secondary contact

Exclusion Criteria:

* currently pregnant or trying to get pregnant;
* plans to move or leave the state during the study, including pending legal action;
* self reported past year suicide attempt or self-reported past year suicidal thoughts with a plan;
* Patient is currently being treated for an acute illness or has a condition that is not stable including but not limited to an upcoming surgical procedure, hospitalization, or complex treatment regimen (e.g., chemotherapy, HCV treatment, has surgery scheduled, has procedures anticipated, has anticipated dose changes with other medication), that is likely to require ongoing, intense clinical management

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-07-25 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Retention in MAT | up to 90 days post randomization
  Proportion of patients attending one or more visits with MAT providers every 30 days for up to 90 days post randomization according to the medical or pharmacy record
Relapse to drug use | up to 90 days post randomization
  Proportion of patients who relapse to drug use, defined as absence of the MAT medication and presence of heroin or other illicit opioids. Measured by toxicological (urine or oral) analysis, with samples collected at every visit (i.e., <every 30 days), or at the 3-month interview at the research site. For patients attending visits, the toxicological results will consider those in the medical or pharmacy record. Urine or oral samples will test for drugs of abuse plus fentanyl, using a rapid qualitative immunoassay.

SECONDARY OUTCOMES:
Primary care visits | up to 90 days post randomization
  Measured by patient self-report, patient medical record review, or by direct contact with the facility, clinician, or both.
  The self report item asks: How many times did you visit your primary care provider (do NOT count visits to providers at the emergency department) in the past 90 DAYS (since starting this study)?
  1. Never, no provider
  2. Never, but I have a provider
  3. Once or twice
  4. 3-5 times
  5. 6 or more times
Emergency department visits | up to 90 days post randomization
  Measured by patient self-report, patient medical record review, or by direct contact with the facility, clinician, or both.
  The self report item asks: How often did you visit the emergency room in the past 90 DAYS (since starting this study)?
  1. Never
  2. Once or twice
  3. 3-5 times
  4. 6 or more times
Hospitalizations | up to 90 days post randomization
  Measured as by patient self-report, patient medical record review, or by direct contact with the facility, clinician, or both.
  The self report item asks: How often were you hospitalized in the past 90 DAYS (since starting this study)?
  1. Never
  2. Once or twice
  3. 3-5 times
  4. 6 or more times

OTHER OUTCOMES:
Engagement in MAT | up to 30 days post randomization
  Proportion of patients with one or more visits during the first 30 days post randomization according to the medical or pharmacy record

CONTACTS AND LOCATIONS:
Overall Officials: Traci C Green, PhD, MSc, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and informed consent form will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available after 50% of the sample recruitment has been reached (n=125)
Access Criteria: Other researchers may request data in writing from the principal investigator

REFERENCES:
- [Derived] Green TC, Serafinski R, Clark SA, Rich JD, Bratberg J. Physician-Delegated Unobserved Induction with Buprenorphine in Pharmacies. N Engl J Med. 2023 Jan 12;388(2):185-186. doi: 10.1056/NEJMc2208055. No abstract available. PMID 36630629